CLINICAL TRIAL: NCT06544733
Title: An Operationally Seamless Phase 2/3, Randomized, Active-Controlled Study Evaluating the Safety and Efficacy of an Oral Weekly Regimen of GS-1720 in Combination With GS-4182 Versus Biktarvy in Virologically Suppressed People With HIV-1
Brief Title: Study of Oral Weekly GS-1720 and GS-4182 Versus Biktarvy in People With HIV-1 Who Are Virologically Suppressed
Acronym: WONDERS1
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-695-6509; 2024-511054-50 (Other: European Medicines Agency)
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: HIV-1-Infection
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Phase 2 (Treatment Group 1, Treatment Group 2, and Extension Phase) arms and Phase 3 Extension Phase arm are open-label; Phase 3 Treatment Group 1 and Phase 3 Treatment Group 2 arms are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 2: GS-1720 + GS-4182 (Treatment Group 1) (Experimental): Participants who have been virologically suppressed on bictegravir/emtricitabine/tenofovir alafenamide (BVY) will switch to GS-1720 (650 mg tablet) and GS-4182 (300 mg tablet) coadministered. Participants will receive a 1-day loading dose of GS-1720 (1300 mg) and GS-4182 (600 mg) on Day 1. Thereafter, participants will take weekly doses of single agent GS-1720 (650 mg) and GS-4182 (300 mg) coadministered for at least 48 weeks.
  Interventions: Drug: GS-1720; Drug: GS-4182
- Phase 2: Bictegravir/emtricitabine/tenofovir alafenamide (BVY) (Treatment Group 2) (Active Comparator): Participants who have been virologically suppressed on bictegravir/emtricitabine/tenofovir alafenamide (BVY) will continue receiving BVY daily for at least 48 weeks.
  Interventions: Drug: Bictegravir/emtricitabine/tenofovir alafenamide
- Phase 2 Extension Phase: GS-1720/GS-4182 Fixed-dose Combination (FDC) (Experimental): At the end of the randomized treatment, Phase 2 participants will be given the option to participate in the Extension Phase. Phase 2 Treatment Group 1 will switch to GS-1720/GS-4182 FDC weekly. Phase 2 Treatment Group 2 will receive a loading dose of GS-1720/GS-4182 FDC on Extension Phase Day 1 then, GS-1720/GS-4182 FDC weekly. Participants who choose to enter the Extension Phase will receive GS-1720/GS-4182 FDC tablets until the product becomes available or until Gilead Sciences elects to discontinue the study, whichever occurs first.
  Interventions: Drug: GS-1720/GS-4182 FDC
- Phase 3: GS-1720/GS-4182 FDC + Placebo to Match (PTM) BVY (Treatment Group 1) (Experimental): Participants who have been virologically suppressed on BVY will switch from BVY to GS-1720/GS-4182 FDC tablets weekly + placebo-to-match (PTM) BVY once daily. In addition, participants will receive a 1-day loading dose regimen of GS-1720/GS-4182 FDC on Day 1.
  Participants will receive treatment for at least 96 weeks.
  Interventions: Drug: Placebo to Match BVY; Drug: GS-1720/GS-4182 FDC
- Phase 3: BVY Placebo to Match GS-1720/GS-4182 FDC + BVY (Treatment Group 2) (Active Comparator): Participants who have been virologically suppressed on BVY will continue receiving oral BVY daily. In addition, participants will receive a 1-day loading dose of PTM GS-1720/GS-4182 on Day 1 and weekly PTM thereafter. Participants will receive treatment for at least 96 weeks.
  Interventions: Drug: Bictegravir/emtricitabine/tenofovir alafenamide; Drug: Placebo to Match GS1720/GS-4182 FDC
- Phase 3 Extension Phase: GS-1720/GS-4182 Fixed-dose Combination (FDC) (Experimental): After the end of blinded treatment, Phase 3 participants will be given the option to participate in the Extension Phase. Phase 3 Treatment Group 1 will switch to GS-1720/GS-4182 FDC weekly. Phase 3 Treatment Group 2 will receive a 1-day loading dose of GS-1720/GS-4182 FDC on Extension Phase Day 1, then GS-1720/GS-4182 FDC weekly. Participants who choose to enter the Extension Phase will receive GS-1720/GS-4182 FDC tablets until the product becomes available or until Gilead Sciences elects to discontinue the study, whichever occurs first.
  Interventions: Drug: GS-1720/GS-4182 FDC

INTERVENTIONS:
Drug: GS-1720 — Tablets administered orally without regard to food
  Arms: Phase 2: GS-1720 + GS-4182 (Treatment Group 1)
Drug: GS-4182 — Tablets administered orally without regard to food
  Arms: Phase 2: GS-1720 + GS-4182 (Treatment Group 1)
Drug: Placebo to Match BVY — Tablets administered orally without regard to food
  Arms: Phase 3: GS-1720/GS-4182 FDC + Placebo to Match (PTM) BVY (Treatment Group 1)
Drug: Bictegravir/emtricitabine/tenofovir alafenamide — Tablets administered orally without regard to food
  Other Names: Biktarvy®
  Arms: Phase 2: Bictegravir/emtricitabine/tenofovir alafenamide (BVY) (Treatment Group 2); Phase 3: BVY Placebo to Match GS-1720/GS-4182 FDC + BVY (Treatment Group 2)
Drug: GS-1720/GS-4182 FDC — Tablets administered orally without regard to food
  Arms: Phase 2 Extension Phase: GS-1720/GS-4182 Fixed-dose Combination (FDC); Phase 3 Extension Phase: GS-1720/GS-4182 Fixed-dose Combination (FDC); Phase 3: GS-1720/GS-4182 FDC + Placebo to Match (PTM) BVY (Treatment Group 1)
Drug: Placebo to Match GS1720/GS-4182 FDC — Tablets administered orally without regard to food
  Arms: Phase 3: BVY Placebo to Match GS-1720/GS-4182 FDC + BVY (Treatment Group 2)

SUMMARY:
The goal of this clinical study is to learn more about the experimental drugs GS-1720 and GS-4182; to compare the combination of GS-1720 and GS-4182 with the current standard-of-care treatment bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF, BVY), to see if the combination of GS-1720 and GS-4182 is safe and if it works for treating human immunodeficiency virus type 1 (HIV-1) infection.

This study has two phases: Phase 2 and Phase 3.

The primary objectives of this study are:

Phase 2: To evaluate the efficacy of switching to oral weekly GS-1720 in combination with GS-4182 versus continuing BVY in virologically suppressed people with HIV-1 (PWH) at Week 24.

Phase 3: To evaluate the efficacy of switching to oral weekly GS-1720/GS-4182 Fixed-dose combination (FDC) tablet regimen versus continuing BVY in virologically suppressed PWH at Week 48.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented plasma HIV-1 RNA < 50 copies/mL for ≥ 24 weeks before and at screening.
* Receiving BVY for ≥ 24 weeks prior to screening.

Key Exclusion Criteria:

* Prior use of, or exposure to LEN, GS-1720, or GS-4182.
* History of virologic failure while on an integrase strand-transfer inhibitor (INSTI)-based regimen.
* Documented integrase strand-transfer inhibitor (INSTI) resistance, specifically, resistance-associated mutations (RAMs) E92G/Q, G118R, F121Y, Y143C/H/R, S147G, Q148H/K/R, N155H/S, or R263K in the integrase gene.
* Prior use of any long-acting (LA) parenteral antiretrovirals (ARV) such as monoclonal antibodies (mAbs) or broadly neutralizing antibodies (bNAbs) targeting HIV-1, injectable cabotegravir (including oral cabotegravir lead-in), or injectable rilpivirine.
* Any of the following laboratory values at screening:

  * Clusters of differentiation 4 (CD4) cell count < 200 cells/mm^3 at screening
  * Glomerular filtration rate < 60 mL/min according to the Modification of Diet in Renal Disease formula
  * Hepatic transaminases (aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 1.5 × upper limit of normal (ULN)
  * Direct bilirubin > 1.5 × ULN
  * Platelets count < 50,000 cells/mm^3
  * Hemoglobin < 8.0 g/dL
* Active or occult hepatitis B virus (HBV) infection.
* Active hepatitis C virus (HCV).

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Proportion of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 24 as Determined by the United States (US) Food and Drug Administration (FDA)-defined Snapshot Algorithm | Week 24
Phase 3: Proportion of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 48 as Determined by the US FDA-defined Snapshot Algorithm | Week 48

SECONDARY OUTCOMES:
Phase 2: Proportion of Participants With HIV-1 RNA ≥ 50 copies/mL at Week 12 as Determined by the US FDA-defined Snapshot Algorithm | Week 12
Phase 2: Proportion of Participants With HIV-1 RNA ≥ 50 copies/mL at Week 48 as Determined by the US FDA-defined Snapshot Algorithm | Week 48
Phase 2: Proportion of Participants With HIV-1 RNA < 50 Copies/mL at Week 12 as Determined by the US FDA-defined Snapshot Algorithm | Week 12
Phase 2: Proportion of Participants With HIV-1 RNA < 50 Copies/mL at Week 24 as Determined by the US FDA-defined Snapshot Algorithm | Week 24
Phase 2: Proportion of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 as Determined by the US FDA-defined Snapshot Algorithm | Week 48
Phase 2: Change From Baseline in Clusters of Differentiation 4 (CD4+) T-cell Count at Week 12 | Baseline, Week 12
Phase 2: Change From Baseline in CD4+ T-cell Count at Week 24 | Baseline, Week 24
Phase 2: Change From Baseline in CD4+ T-cell Count at Week 48 | Baseline, Week 48
Phase 2: Percentage of Participants Experiencing Treatment Emergent Adverse Events (TEAEs) Through Week 12 | First dose date up to Week 12
Phase 2: Percentage of Participants Experiencing TEAEs Through Week 24 | First dose date up to Week 24
Phase 2: Percentage of Participants Experiencing TEAEs Through Week 48 | First dose date up to Week 48
Phase 2: Percentage of Participants Experiencing Treatment-emergent Laboratory Abnormalities Through Week 12 | First dose date up to Week 12
Phase 2: Percentage of Participants Experiencing Treatment-emergent Laboratory Abnormalities Through Week 24 | First dose date up to Week 24
Phase 2: Percentage of Participants Experiencing Treatment-emergent Laboratory Abnormalities Through Week 48 | First dose date up to Week 48
Phase 2: Pharmacokinetic (PK) Parameter: Cmax of GS-1720 and Lenacapavir (LEN) | Day 1 up to Week 48
  Cmax is defined as the maximum observed concentration of drug.
Phase 2: PK Parameter: Tmax of GS-1720 and LEN | Day 1 up to Week 48
  Tmax is defined as the time (observed time point) of Cmax.
Phase 2: PK Parameter: Ctau of GS-1720 and LEN | Day 1 up to Week 48
  Ctau is defined as the observed drug concentration at the end of the dosing interval.
Phase 2: PK Parameter: AUCtau of GS-1720 and LEN | Day 1 up to Week 48
  AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Phase 3: Proportion of Participants With HIV-1 RNA ≥ 50 copies/mL at Week 96 as Determined by the US FDA-defined Snapshot Algorithm | Week 96
Phase 3: Proportion of Participants With HIV-1 RNA < 50 copies/mL at Week 48 as Determined by the US FDA-defined Snapshot Algorithm | Week 48
Phase 3: Proportion of Participants With HIV-1 RNA < 50 copies/mL at Week 96 as Determined by the US FDA-defined Snapshot Algorithm | Week 96
Phase 3: Change From Baseline in CD4+ T-cell Count at Week 48 | Baseline, Week 48
Phase 3: Change From Baseline in CD4+ T-cell Count at Week 96 | Baseline, Week 96
Phase 3: Percentage of Participants Experiencing TEAEs Through Week 48 | First dose date up to Week 48
Phase 3: Proportion of Participants Experiencing TEAEs Through Week 96 | First dose date up to Week 96
Phase 3: Percentage of Participants Experiencing Treatment-emergent Laboratory Abnormalities Through Week 48 | First dose date up to Week 48
Phase 3: Percentage of Participants Experiencing Treatment-emergent Laboratory Abnormalities Through Week 96 | First dose date up to Week 96

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (39):
- United States (35):
  - UAB 1917 Research Clinic, Birmingham, Alabama
  - Pacific Oaks Medical Group, Beverly Hills, California
  - Ruane Clinical Research Group, Los Angeles, California
  - Mills Clinical Research, Los Angeles, California
  - BIOS Clinical Research, Palm Springs, California
  - UCSF Division of HIV, Infectious Diseases & Global Medicine, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Midland Florida Clinical Research Center, LLC, DeLand, Florida
  - CAN Community Health, Fort Lauderdale, Florida
  - Midway and Immunology Research Center, Ft. Pierce, Florida
  - AIDS Healthcare Foundation - The Kinder Medical Group, Miami, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - Orlando Immunology Center, Orlando, Florida
  - CAN Community Health, Sarasota, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - Metro Infectious Disease Consultants, P.L.L.C., Decatur, Georgia
  - Mercer University, Department of Internal Medicine, Macon, Georgia
  - Chatham County Health Department, Savannah, Georgia
  - Be Well Medical Center, Berkley, Michigan
  - KC CARE Health Center, Kansas City, Missouri
  - Saint Michael's Medical Center, Newark, New Jersey
  - AXCES Research Group, LLC, Santa Fe, New Mexico
  - NewYork-Presbyterian Queens, Flushing, New York
  - NYU Langone Health Vaccine Center, New York, New York
  - Rosedale Health and Wellness, Huntersville, North Carolina
  - Central Texas Clinical Research, Austin, Texas
  - St Hope Foundation, Inc., Bellaire, Texas
  - Prism Health North Texas, Oak Cliff Health Center, Dallas, Texas
  - North Texas Infectious Diseases Consultants, PA, Dallas, Texas
  - AXCES Research Group, LLC, El Paso, Texas
  - Texas Centers for Infectious Disease Associates, Fort Worth, Texas
  - The Crofoot Research Center, INC., Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Peter Shalit, MD, Seattle, Washington
- Puerto Rico (4):
  - Centro Ararat, Inc., San Juan, PR
  - Clinical Research Puerto Rico, San Juan, PR
  - HOPE Clinical Research, San Juan, PR
  - Proyecto ACTC, San Juan, PR

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06544733